CLINICAL TRIAL: NCT02278211
Title: Prediction of Recurrent Events With 18F-Fluoride to Identify Ruptured and High-risk Coronary Artery Plaques in Patients With Myocardial Infarction
Brief Title: Prediction of Recurrent Events With 18F-Fluoride
Acronym: PREFFIR
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Oxford University Hospitals NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); NHS Grampian (Other Government); Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PREFFIR
Record Dates: First submitted 2014-10-15; First posted 2014-10-29 (Estimated); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low Coronary Atherosclerotic Plaque Activity: Patients hospitalised with myocardial infarction and angiographically proven multivessel coronary artery disease found to have Low Coronary Atherosclerotic Plaque Activity in PET CT scan
- High Coronary Atherosclerotic Plaque Activity: Patients hospitalised with myocardial infarction and angiographically proven multivessel coronary artery disease found to have High Coronary Atherosclerotic Plaque Activity in PET CT scan

SUMMARY:
This is a multi-centre observational study. It will make use of the positron emission tomography (PET) tracer 18F-sodium fluoride (18F-NaF) as a marker of coronary plaque vulnerability to detect culprit and non-culprit unstable coronary plaques in patients with recent myocardial infarctions. The investigators will then perform long-term follow-up of these patients to determine the prognostic significance of coronary 18F-NaF uptake

DETAILED DESCRIPTION:
The investigators intend to recruit 700 patients hospitalised with myocardial infarction and proven multivessel coronary artery disease. All patients will undergo a combined CT coronary angiogram (CTCA) and PET scan using 18F-NaF as a tracer. Patients will then have clinical follow-up before undergoing a repeat CTCA at 2 years to assess progression of coronary disease. Clinical review of all patients will continue until study completion (given 2 years of recruitment this is likely to last 4 years) and following this the investigators will continue to monitor for further cardiovascular events via review of patient electronic health records for a further 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥50 years with recent (<21 days) type 1 myocardial infarction and angiographically proven multi-vessel coronary artery disease defined as at least two major epicardial vessels with any combination of either (a) >50% luminal stenosis, or (b) previous revascularization (percutaneous coronary intervention or coronary artery bypass graft surgery).
2. Provision of informed consent prior to any study specific procedures

Exclusion Criteria:

1. Inability or unwilling to give informed consent
2. Women who are pregnant, breastfeeding or of child-bearing potential (women who have experienced menarche, are pre-menopausal and have not been sterilised) will not be enrolled into the trial
3. Major intercurrent illness with life expectancy <2 year
4. Renal dysfunction (estimated glomerular filtration rate ≤30 mL/min/1.73 m2)
5. Contraindication to iodinated contrast agent, positron emission tomography or computed tomography
6. Atrial fibrillation
7. Previous recruitment into the trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent (<21 days) type 1 myocardial infarction and multi-vessel coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 995 (Actual)
Dates: Start 2015-10; Primary Completion 2022-03 (Actual); Study Completion 2022-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Newby, PhD, Study Director — University of Edinburgh
Locations (1):
- Edinburgh Heart Centre, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Background] Joshi NV, Vesey AT, Williams MC, Shah AS, Calvert PA, Craighead FH, Yeoh SE, Wallace W, Salter D, Fletcher AM, van Beek EJ, Flapan AD, Uren NG, Behan MW, Cruden NL, Mills NL, Fox KA, Rudd JH, Dweck MR, Newby DE. 18F-fluoride positron emission tomography for identification of ruptured and high-risk coronary atherosclerotic plaques: a prospective clinical trial. Lancet. 2014 Feb 22;383(9918):705-13. doi: 10.1016/S0140-6736(13)61754-7. Epub 2013 Nov 11. PMID 24224999
- [Background] Dweck MR, Chow MW, Joshi NV, Williams MC, Jones C, Fletcher AM, Richardson H, White A, McKillop G, van Beek EJ, Boon NA, Rudd JH, Newby DE. Coronary arterial 18F-sodium fluoride uptake: a novel marker of plaque biology. J Am Coll Cardiol. 2012 Apr 24;59(17):1539-48. doi: 10.1016/j.jacc.2011.12.037. PMID 22516444
- [Background] Mohler ER 3rd, Alavi A, Wilensky RL. (18)F-fluoride imaging for atherosclerosis. J Am Coll Cardiol. 2012 Oct 23;60(17):1711-2; author reply p.1712-3. doi: 10.1016/j.jacc.2012.06.038. No abstract available. PMID 23079119
- [Background] Derlin T, Toth Z, Papp L, Wisotzki C, Apostolova I, Habermann CR, Mester J, Klutmann S. Correlation of inflammation assessed by 18F-FDG PET, active mineral deposition assessed by 18F-fluoride PET, and vascular calcification in atherosclerotic plaque: a dual-tracer PET/CT study. J Nucl Med. 2011 Jul;52(7):1020-7. doi: 10.2967/jnumed.111.087452. Epub 2011 Jun 16. PMID 21680686
- [Background] Derlin T, Richter U, Bannas P, Begemann P, Buchert R, Mester J, Klutmann S. Feasibility of 18F-sodium fluoride PET/CT for imaging of atherosclerotic plaque. J Nucl Med. 2010 Jun;51(6):862-5. doi: 10.2967/jnumed.110.076471. Epub 2010 May 19. PMID 20484438
- [Derived] Moss AJ, Doris MK, Andrews JPM, Bing R, Daghem M, van Beek EJR, Forsyth L, Shah ASV, Williams MC, Sellers S, Leipsic J, Dweck MR, Parker RA, Newby DE, Adamson PD. Molecular Coronary Plaque Imaging Using 18F-Fluoride. Circ Cardiovasc Imaging. 2019 Aug;12(8):e008574. doi: 10.1161/CIRCIMAGING.118.008574. Epub 2019 Aug 6. PMID 31382765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start date- September 2015 Recruitment end date - February 2020 The study was conducted in 9 centres across 4 countries (Scotland, England, United States and Australia) [Note groups combined in below as participants only allocated to group after PET CT Scan analysed. Unable to report on reason not completed separately. as scan not complete at this point]
Pre-assignment Details: After consent 283 participants were excluded reasons below:
  Changed mind (n=142) Unable to scan within protocol window (n=82) Health subsequently deteriorated precluding inclusion (n=22) Unable to contact patient (n=19) Ineligible (n=10) Deceased (n=6) Clinician/investigator decision (n=2) 6 Participants attended baseline but did not complete the PET-CT Scan- were not allocated an arm. Reasons below: Claustrophobia (n=3) Panic attack (n=1) Anxious (n=1) Scanner malfunction (n=1)
Groups:
- Study Cohort: Patients hospitalised with myocardial infarction and angiographically proven multivessel coronary artery disease
Period: Overall Study
Arm/Group | Study Cohort
Started | 706
Completed | 704
Not Completed | 2
Not completed — Unable to analyse PET scan | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics split into low or high atherosclerotic plaque activity assessed after CT PET scan.
Groups:
- Low Coronary Atherosclerotic Plaque Activity: Low coronary atherosclerotic plaque activity
- High Coronary Atherosclerotic Plaque Activity: High coronary atherosclerotic plaque activity
- Total: Total of all reporting groups
Arm/Group | Low Coronary Atherosclerotic Plaque Activity | High Coronary Atherosclerotic Plaque Activity | Total
Number analyzed (Participants) | 283 | 421 | 704
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (7.4) | 65.1 (8.4) | 63.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 42 | 103
  Male | 222 | 379 | 601
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass index [Mean (Standard Deviation); unit: kg/m2] | 28.6 (4.7) | 28.1 (4.2) | 28.3 (4.4)
Smoking status [Count of Participants; unit: Participants]
  Current | 90 | 103 | 193
  Former | 91 | 134 | 225
  Never | 102 | 184 | 286
Hypertension [Count of Participants; unit: Participants] | 119 | 232 | 351
Hypercholesterolemia [Count of Participants; unit: Participants] | 162 | 236 | 398
Diabetes [Count of Participants; unit: Participants] | 40 | 78 | 118
Coronary artery disease [Count of Participants; unit: Participants] | 41 | 98 | 139
Myocardial infarction [Count of Participants; unit: Participants] | 36 | 66 | 102
Percutaneous coronary intervention [Count of Participants; unit: Participants] | 28 | 72 | 100
Coronary artery bypass graft surgery [Count of Participants; unit: Participants] | 12 | 19 | 31
Peripheral vascular disease [Count of Participants; unit: Participants] | 12 | 9 | 21
Cerebrovascular disease [Count of Participants; unit: Participants] | 10 | 23 | 33
Electrocardiography findings [Count of Participants; unit: Participants]
  ST-segment elevation myocardial infarction | 189 | 274 | 463
  Non-ST-segment elevation myocardial infarction | 94 | 145 | 239
  Missing data points | 0 | 2 | 2
GRACE score [Mean (Standard Deviation); unit: scores on a scale] — The Global Registry of Acute Coronary Events - a guideline-recommended risk stratification tool for patients presenting with acute coronary syndromes. A GRACE score of 141-372 is considered high risk, while a score of 1-108 is considered low risk. A score of 109-140 is considered intermediate risk. The odds of in-hospital mortality increase significantly with a higher GRACE score.
  scores on a scale | 113 (22) | 121 (26) | 118 (25)
Severity of obstructive coronary artery disease [Count of Participants; unit: Participants]
  1 Vessel | 12 | 16 | 28
  2 Vessels | 163 | 224 | 387
  3 Vessels | 90 | 149 | 239
  Left main stem disease | 18 | 32 | 50
Percutaneous coronary intervention [Count of Participants; unit: Participants] | 267 | 404 | 671
Medication [Count of Participants; unit: Participants]
  Aspirin: Yes | 268 | 405 | 673
  Aspirin: No | 15 | 16 | 31
  P2Y12 receptor antagonist: Yes | 279 | 409 | 688
  P2Y12 receptor antagonist: No | 4 | 12 | 16
  Anticoagulant therapy: Yes | 17 | 25 | 42
  Anticoagulant therapy: No | 266 | 396 | 662
  Statin: Yes | 260 | 393 | 653
  Statin: No | 23 | 28 | 51
  ACE inhibitor or ARB: Yes | 250 | 373 | 623
  ACE inhibitor or ARB: No | 33 | 48 | 81
  β-Adrenergic receptor antagonist: Yes | 233 | 340 | 573
  β-Adrenergic receptor antagonist: No | 50 | 81 | 131
  Calcium-channel antagonist: Yes | 19 | 45 | 64
  Calcium-channel antagonist: No | 264 | 376 | 640
  Nitrate: Yes | 158 | 226 | 384
  Nitrate: No | 125 | 195 | 320
  Other antianginal therapy: Yes | 8 | 14 | 22
  Other antianginal therapy: No | 275 | 407 | 682
  Mineralocorticoid receptor antagonist: Yes | 21 | 21 | 42
  Mineralocorticoid receptor antagonist: No | 262 | 400 | 662
  Other diuretic therapy: Yes | 22 | 32 | 54
  Other diuretic therapy: No | 261 | 389 | 650

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Death, Non-fatal Recurrent Myocardial Infarction or Unscheduled Coronary Revascularisation
Description: To determine whether coronary 18F-fluoride uptake is associated with major adverse cardiac events in patients with multi-vessel coronary artery disease and recent myocardial infarction. Participants were followed up by site investigators until the last recruited patient had completed their 2-year follow-up visit.
Time Frame: 2 years
Population: Clinical follow-up was available for all study participants. At study completion, follow-up was available for 693 participants (98.4%). Over a median of 4 years (IQR, 3-5 years), there were 2582 patient-years of follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Coronary Atherosclerotic Plaque Activity | High Coronary Atherosclerotic Plaque Activity
Number analyzed (Participants) | 283 | 421
Participants | 51 | 90
Statistical Analysis 1: Comparison: Low Coronary Atherosclerotic Plaque Activity vs High Coronary Atherosclerotic Plaque Activity; Test type: Other; p = 0.20, Log Rank; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.89 to 1.76]

2. Secondary Outcome: All Cause Death
Description: All cause death. Participants were followed up by site investigators until the last recruited patient had completed their 2-year follow-up visit.
Time Frame: 2 years
Population: All cause death
Measure: Count of Participants; unit: Participants
Arm/Group | Low Coronary Atherosclerotic Plaque Activity | High Coronary Atherosclerotic Plaque Activity
Number analyzed (Participants) | 283 | 421
Participants | 9 | 30
Statistical Analysis 1: Comparison: Low Coronary Atherosclerotic Plaque Activity vs High Coronary Atherosclerotic Plaque Activity; Test type: Other; p = 0.02, Log Rank; Hazard Ratio (HR) = 2.43, 95% CI 2-sided [1.15 to 5.12]

3. Secondary Outcome: Each Individual Component End-point of the Composite End-point of Major Adverse Cardiac Event
Description: Cardiac death, Nonfatal myocardial infarction, Unscheduled coronary revascularization
Time Frame: 2 years
Population: Cardiac death, Nonfatal myocardial infarction, Unscheduled coronary revascularization
Measure: Count of Participants; unit: Participants
Arm/Group | Low Coronary Atherosclerotic Plaque Activity | High Coronary Atherosclerotic Plaque Activity
Number analyzed (Participants) | 55 | 98
Participants
  Cardiac death | 2 | 10
  Nonfatal myocardial infarction | 17 | 37
  Unscheduled coronary revascularization | 36 | 51

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored for up to 2 years; serious and/or other adverse events were assessed up to 48 hours post PET CT scan
Description: Adverse events were collected irrespective of plaque activity status and therefore cannot be separated. Adverse events were not assessed per group/arm.
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 39/704
Serious Adverse Events (participants affected / at risk) | 2/704
Other Adverse Events (participants affected / at risk) | 13/704
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Cohort (N=704)
Beta-blocker induced bradycardia (Cardiac disorders) | 1 (1) — Admitted with heart failure to CCU, exacerbated by beta blocker
Palpitations (Cardiac disorders) | 1 (1) — Subject admitted to hospital with palpitations following caffeine intake
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Cohort (N=704)
Contrast reaction (Skin and subcutaneous tissue disorders) | 8 (8) — Contrast reaction
Cannula access site (Product Issues) | 5 (5) — Cannula access site

LIMITATIONS AND CAVEATS:
We had a lower than anticipated event rate in the study population. This led us to change our primary end point to include unscheduled coronary revascularization. Our study was a longitudinal cohort study, we could only assess associations rather than causality. Low inclusion of women, reflects the lower proportion of women who present with ST-segment elevation MI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is agreed that the Co-Sponsors shall publish the results of the full Study and that the Site and the Site Principal Investigator shall not publish the results of the Study carried out at the Site without the prior permission in writing from Edinburgh (which shall not be unreasonably withheld) and in any case not prior to the publication of the results of the full Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT02278211/Prot_SAP_000.pdf